CLINICAL TRIAL: NCT01001273
Title: Hyperinsulinemic Normoglycemic Clamp for Pancreas and Simultaneous Pancreas/Kidney Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Dr Steven Paraskevas & Dr Mazen Hassanain, MUHC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SDR-09-061
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Postoperative Complications
Keywords: Pancreas Transplantation; Kidney Transplantation; Organ Transplantation; Pancreas and Simultaneous Pancreas/Kidney Transplant Recipients
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): Hyperinsulinemic Normoglycemic Clamp will be started at the time of surgery (before incision) and will be continue for 3 days.
  Interventions: Other: Hyperinsulinemic Normoglycemic Clamp
- Control Group (No Intervention): Patients in the control group will receive standard care.

INTERVENTIONS:
Other: Hyperinsulinemic Normoglycemic Clamp — The patient receives insulin intravenous infusion at 2ml units/kg/min. Dextrose 20% (D20W ®) will be titrated to maintain blood glucose between 4 - 6 mmol/L (72 - 108 mg/dl).
  Arms: Study Group

SUMMARY:
This study proposes a simple and safe way of lowering this complicate rate, while improving graft recovering and protecting the graft as it recovers from the transplant. The investigators hypothesize that by maintaining a tight glucose control via a glucose-insulin clamp during surgery and 72 hours post-operatively the investigators will be able to lower the complication rate by 50%.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient over 18 years of age
* Patient is about to receive a pancreas or a simultaneous pancreas/kidney transplant
* Able to give written informed consent prior to any study specific procedure

Exclusion Criteria:

* Multi-organ transplant other than kidney transplant
* No central venous access available to deliver the D20W solution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
The number of post-transplants all complications up to 30 days (Clavien grading). | 30 days post-operative

SECONDARY OUTCOMES:
The number of 30 days post-transplant serious medical complication (Clavien grade 3, 4) | 30 days post-op
The length of hospital stay (days) | Length of hospital stay (day 1 until discharge)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Royal Victoria, Montreal, Quebec, Canada